CLINICAL TRIAL: NCT02393300
Title: Comparison of Topical Versus Intravenous Tranexamic Acid in Primary Total Knee Arthroplasty：A Prospective Randomized Study
Brief Title: Comparison of Topical Versus Intravenous Tranexamic Acid in TKA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, zhoukaidi, MD in Shanghai Jiao Tong University School of Medicine, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: JTU-GK-011
Record Dates: First submitted 2015-03-15; First posted 2015-03-19 (Estimated); Last update posted 2018-04-04 (Actual); Status verified 2015-11

CONDITIONS: Total Blood Loss
Keywords: tranexamic acid; blood loss; topical administration; intravenous administration
MeSH Terms: conditions — Exsanguination; Hemorrhage | interventions — Saline Solution; Sodium Chloride; Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group1 (Placebo Comparator): 60 Milliliters（ml）Normal saline (0.9% sodium chloride) will be applied by soaking the knee cavity for at least 3 minutes before wound closure and then sucked away.
  Interventions: Drug: normal saline
- Group2 (Experimental): two-dose intravenous tranexamic acid will be applied as follow: 10mg/kg of Tranexamic Acid in 100 Milliliters（ml) normal saline (0.9% sodium chloride),the first dose 15' before the tourniquet deflation and the second dose at 180' after the first dosage
  Interventions: Drug: Tranexamic Acid
- Group 3 (Experimental): 3g Tranexamic Acid diluted to 60 Milliliters（ml） with normal saline (0.9% sodium chloride) will be applied by soaking the knee cavity for at least 3 minutes before wound closure and then sucked away.
  Interventions: Drug: Tranexamic Acid

INTERVENTIONS:
Drug: normal saline — The normal saline solution will be prepared under sterile conditions. In the operation room the sterile bag containing the solution will be given to the scrub nurse. The contents (60 ml) will be emptied in a sterile surgical bowl and the nurse will ask the surgeon to apply the solution before wound closure.The dosage and applying route can also be looked up in doctor's order sheet.
  Other Names: 0.9% sodium chloride
  Arms: Group1
Drug: Tranexamic Acid — The Tranexamic Acid solution will be prepared under sterile conditions. In the operation room the sterile bag containing the solution will be given to the scrub nurse. The contents (60 ml) will be emptied in a sterile surgical bowl and the nurse will ask the surgeon to apply the solution before wound closure.The dosage and applying route can also be looked up in doctor's order sheet.
  Other Names: Cyclokapron
  Arms: Group 3
Drug: Tranexamic Acid — The Tranexamic Acid solution will be prepared under sterile conditions. In the operation room the sterile bag containing the solution will be given to the circuit nurse and the circuit nurse will ask the anesthetist to apply the solution intravenously before tourniquet deflation. The dosage and applying route can also be looked up in doctor's order sheet.
  Other Names: Cyclokapron
  Arms: Group2

SUMMARY:
Previous studies in both the cardiovascular and orthopedic study have shown tranexamic acid (TXA) reduces blood loss and post-operative blood transfusion rate largely without major complications . In addition, many meta-analyses have confirmed these results . However, there is little information about comparison among the different routes of TXA administration in TKA. Therefore, this study has been designed to determine which administration route of TXA is more effective and safety.

DETAILED DESCRIPTION:
Objectives:To assess the efficacy and safety between the two different applying routes.

Patients in this project will be randomly divided into three groups , one group is a blank group and the rest two receive either the topical or the intravenous form of tranexamic acid during unilateral TKA(total knee arthroplasty).The total blood loss(TBL) will be calculated as the primary outcome for efficacy while Deep Vein Thrombosis、Pulmonary Embolism、Acute Myocardial Infarction 、 Acute Kidney Infarction and Cerebral Infarction events will be recorded to assess the safety of the tranexamic acid during a six-week follow-up for each patient.

All surgery are under general anesthesia, through direct lateral approach with cementless prosthesis.For all patients, the drain tube will be clamped and closed completely for 2 hours; then the clamp will be fully opened.

ELIGIBILITY:
Inclusion Criteria:

1. Consented to join in our project.
2. Adult patients (greater than 18 years old)
3. Patients scheduled for primary unilateral knee arthroplasty

Exclusion Criteria:

1. Patients who refuse to sign the Inform Consent
2. Had an allergy to TXA.
3. Using anticoagulant drugs within a week.
4. Coagulopathy (preoperative platelet count <150,000/mm3,International Sensitivity Index（INR）>1.4, prolonged Activated Partial Thromboplastin Time，Prothrombin Time ，or thrombin time >1.4 times longer than normal.
5. Breastfeeding
6. Major comorbidities: Severe ischemic heart disease(class III and IV of New York Heart Association); sleep apnea syndrome; renal dysfunction ( glomerular filtration rate<60); or hepatic disfunction(glutamic-pyruvic transaminase>80 or glutamic oxalacetic transaminase>80).Retinopathy (disturbances of color vision).

9.History of thromboembolic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2015-05 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Total Blood Loss（TBL） | calculated by an equation at the fifth postoperative day
  Total Blood Loss（TBL） was calculated with equations described by Gross et al.

SECONDARY OUTCOMES:
Transfusion rates | from the day of surgery to the day of discharge,an expected average of 7 days
  Include The number of units of perioperative blood transfusions, both intraoperative and postoperative, over the course of the patient's hospital stay

OTHER OUTCOMES:
Venous thromboembolic event (symptomatic deep vein thrombosis or pulmonary | twelve weeks after surgery
  Clinically proven symptomatic deep vein thrombosis (DVT) or pulmonary embolism
other thromboembolic event | twelve weeks after surgery
  Clinically proven Acute Myocardial Infarction、acute kidney infarction or cerebral infarction
drainage output | it will be recorded at the first day and the second day after surgery
human serum albumin usage | from the day of surgery to the day of discharge,an expected average of 7 days
  the investigators will record the dosage of the human blood albumin used in each patient.
American Society of Anesthesiologists Physical Status Classification (ASA class) | at the day of surgery
Disseminated Intravascular Coagulation（DIC） | at any day before surgery and the first the fifth day after surgery

CONTACTS AND LOCATIONS:
Overall Officials: jianmin feng, master, Principal Investigator — ruijin hospital，shanghai
Locations (1):
- Orthopedic Department of Ruijin hospital, Shanghai, Shanghai Municipality, China